CLINICAL TRIAL: NCT07137117
Title: The Effect of Tele-Counseling Service on Nutrition, Exercise Attitude, and Medication Adherence After Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cansel Bozer, PhD student, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-SBF-CB-04
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Bariatric Surgery (Sleeve Gastrectomy )
Keywords: bariatric surgery; teleconsulting; medication compliance; nutrition exercise attitude
MeSH Terms: conditions — Medication Adherence | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: 2 groups, control and intervention group
Who Masked: Participant, Outcomes Assessor
Masking Description: Teleconsultation services will be provided to the intervention group, which will call them at regular intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Patients in the experimental group will be administered a "Patient Information Form" on the morning of surgery. Standard discharge education will be provided within 72 hours after surgery. After discharge, patients will be contacted at 1, 2, 3 weeks, and 2, 4, and 5 months for informational purposes only; no scales will be administered. During this period, regular follow-up and support will be provided to enhance patient compliance with post-surgical care. The "Interview Information Collection Form" will be used during telephone interviews with patients to collect and evaluate current health data. This practice will ensure the systematic and accurate recording of patients' current conditions. Patients will be contacted at 1, 3, and 6 months to complete the "Medication Adherence Scale" and the "Nutrition and Exercise Attitude Scale," which will collect data on medication adherence and behavioral attitudes.
  Interventions: Other: Behavioral Treatment
- no intervention group (No Intervention): Patients in the control group will be administered a "Patient Information Form" on the morning of surgery. This form will be used to assess the patients' demographic and clinical characteristics. Patients will receive standard discharge education within 72 hours after surgery and then be discharged. Post-discharge follow-up will be conducted via telephone at 1, 3, and 6 months. An "Interview Information Collection Form" will be used during telephone interviews to collect and evaluate current health data. This practice will ensure systematic and accurate recording of patients' current conditions. At each follow-up interview, patients will be administered the "Medication Adherence Scale" and the "Nutrition and Exercise Attitude Scale" to collect data on medication adherence and nutritional and exercise habits. These measurement tools will be used systematically to assess patients' treatment adherence and behavioral attitudes.

INTERVENTIONS:
Other: Behavioral Treatment — Patients in the experimental group will be administered a "Patient Information Form" on the morning of surgery. Standard discharge education will be provided within 72 hours after surgery. After discharge, patients will be contacted at 1, 2, 3 weeks, and 2, 4, and 5 months for informational purposes only; no assessment will be administered. During this period, regular follow-up and support will be provided to enhance patient compliance with post-surgical care. The "Interview Information Collection Form" will be used during telephone interviews with patients to collect and evaluate current health data. This practice will ensure systematic and accurate recording of patients' current conditions. Patients will be contacted at 1, 3, and 6 months to complete the "Medication Adherence Scale" and the "Nutrition and Exercise Attitude Scale," collecting data on medication adherence and behavioral attitudes. These assessments will be used as a systematic approach to monitoring patient adherence t
  Arms: intervention group

SUMMARY:
The aim of this study was to evaluate the effects of teleconsultation service on nutrition, exercise attitudes and medication adherence after bariatric surgery.

DETAILED DESCRIPTION:
Laparoscopic bariatric surgery is a popular procedure that offers proven long-term results in improving obesity-related comorbidities. However, after surgery, patients often experience behavioral adjustments, such as diet, physical activity, and medication use. These adjustments can lead to complications.In particular, poor adherence to vitamin supplements can lead to nutritional deficiencies and related health problems. Lack of adherence to physical activity is also frequently observed. Making lifestyle changes after bariatric surgery is important, and telecounseling stands out as an effective tool in this process. Telecounseling can help patients develop healthy lifestyle habits and increase access to healthcare.Studies show that telephone follow-up and counseling provided via mobile apps after bariatric surgery improves patient health management and treatment adherence. Furthermore, due to the limitations of written educational materials, telephone counseling fosters stronger patient motivation. This method can be customized to individual health needs and facilitates access to healthcare by eliminating geographic limitations. In conclusion, one-on-one telephone counseling can help patients maintain healthy lifestyles after bariatric surgery, improving treatment outcomes and positively impacting long-term health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone laparoscopic bariatric surgery (sleeve gastrectomy only) for the first time,
* Are between the ages of 18 and 65,
* Are conscious and oriented to person, time, and place,
* Can speak Turkish,
* Have no auditory or visual impairments,
* Can use a telephone will be included in the study.

Exclusion Criteria:

* Patients who developed early postoperative complications (bleeding, anastomotic leakage, etc.), were hospitalized for revision surgery, and did not consent to the study will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Reporting Scale | 6 months
  The Medication Adherence Reporting Scale (IAS) is a scale developed to assess medication adherence. The scale asks participants to evaluate five statements based on their own circumstances. This structure allows for the systematic examination of individual attitudes and behaviors toward medication use. The Medication Adherence Reporting Scale (IAS) is assessed using a 5-point Likert-type rating system, with response options of 5=never, 4=rarely, 3=sometimes, 2=often, and 1=very often. The test score is calculated by summing the scores obtained from the scale items.
The Nutrition and Exercise Attitude Scale (NUAS) | 6 months
  The Nutrition and Exercise Attitude Scale (NUAS) was developed in Turkey to measure individuals' attitudes toward nutrition and exercise. Its validity and reliability study was conducted by Yurt (2008). It is structured as a Likert-type scale. This allows individuals to evaluate their own attitudes and behaviors based on various statements. The statements in the scale are rated on a scale according to individuals' level of agreement. Each item in the scale is scored, and a total score is calculated for the subdimensions. Higher scores indicate a more positive attitude in the relevant subdimension. Lower scores indicate that the individual is experiencing difficulties in a particular area. The internal consistency of the scale was assessed using Cronbach's Alpha coefficient and was found to be 0.70. This value indicates that the scale has an acceptable level of internal consistency (Yurt, 2008; Ekici and Yıldız 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Cansel Bozer Uludağ, expert, Principal Investigator
Locations (1):
- Adana City Training and Research Hospital, Adana, Yüreğir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No